CLINICAL TRIAL: NCT02789878
Title: Phase II Study of Neoadjuvant Androgen Deprivation Therapy Plus Abiraterone With or Without Apalutamide for Patients With High-Risk Localized Prostate Cancer Prior to Radical Prostatectomy
Brief Title: Neoadjuvant Androgen Deprivation Therapy Plus Abiraterone With or Without Apalutamide for High-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP 779/15
Record Dates: First submitted 2016-05-25; First posted 2016-06-03 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: Neoadjuvant therapy; High-risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Prednisone; abiraterone; Abiraterone Acetate; apalutamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT and Abiraterone (Experimental): * Goserelin 10.8 mg, single dose, subcutaneously.
  * Abiraterone 1,000 mg, once daily, orally for 3 months.
  * Prednisone 5 mg, once daily, orally for 3 months.
  Interventions: Drug: Goserelin; Drug: Prednisone; Drug: Abiraterone
- ADT, Abiraterone and Apalutamide (Experimental): * Goserelin 10.8 mg, single dose, subcutaneously.
  * Abiraterone 1,000 mg, once daily, orally for 3 months.
  * Prednisone 5 mg, once daily, orally for 3 months.
  * Apalutamide 240 mg, once daily, orally for 3 months.
  Interventions: Drug: Goserelin; Drug: Prednisone; Drug: Abiraterone; Drug: Apalutamide

INTERVENTIONS:
Drug: Goserelin — Androgen Deprivation Therapy
  Other Names: ADT
Drug: Prednisone — Corticosteroid
Drug: Abiraterone — CYP17 inhibitor
  Other Names: Zytiga
Drug: Apalutamide — Androgen-receptor antagonist
  Other Names: ARN-509
  Arms: ADT, Abiraterone and Apalutamide

SUMMARY:
This is a randomized study to evaluate the efficacy and safety neoadjuvant androgen deprivation therapy with goserelin and abiraterone with or without apalutamide prior to radical prostatectomy for patients diagnosed with localized high-risk prostate cancer.

DETAILED DESCRIPTION:
In the prostate specific antigen (PSA) era, about 15% to 20% of patients are diagnosed with high-risk localized disease and radical prostatectomy is a standard therapy for this subgroup of patients. However, despite best local therapy, about 30-60% of high-risk patients will eventually develop biochemical relapse and a significant proportion of these patients may progress with metastatic disease and die from prostate cancer. Currently, there is no data supporting the use of neoadjuvant therapy for patients with high-risk disease since studies failed to demonstrate clinically significant benefit with standard androgen deprivation therapy (ADT). Following improved outcomes in other malignancies with the use of neoadjuvant therapy with active drugs in the metastatic setting, there is a growing interest in evaluating new-generation androgen receptor (AR)-targeted therapy in earlier stages of prostate cancer. Therefore, the goal of this study is to evaluate the efficacy and safety of neoadjuvant therapy with ADT and abiraterone versus maximal androgen blockade using ADT, abiraterone and apalutamide for patients with high-risk localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed prostatic adenocarcinoma
* Non-castrate levels of testosterone (> 150 ng/dL)
* High-risk localized prostate cancer, defined by either:

  * Tumor stage T3 by digital rectal examination, or
  * Primary tumor Gleason score ≥ 8, or
  * PSA ≥ 20 ng/mL
* Willing to undergo prostatectomy as primary treatment for localized prostate cancer
* Adequate hematologic, renal and hepatic function:

  * WBC > 3000/uL
  * Platelets > 150,000/uL
  * Creatinine < 2 mg/dL
  * Bilirubin < 1.5 x upper limit of normal (ULN)
  * AST/ALT < 2 x ULN
* Karnofsky Performance Status (KPS) ≥ 80%
* Able to swallow the study drugs whole as tablets

Exclusion Criteria:

* Pathological finding consistent with small cell, ductal or neuroendocrine carcinoma of the prostate
* Current or prior hormonal therapy, radiation therapy or chemotherapy for prostate cancer
* Evidence of metastatic disease (M1) on imaging studies
* Other prior malignancy less than or equal to 5 years prior to randomization with the exception of squamous or basal cell skin carcinoma
* Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure
* History of prior cardiac arrhythmia.
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Pathologic response | 3 months
  To compare the rate of pathologic complete response (pCR) or pathologic near complete response (pnCR), defined as less than 0,5 cm of residual tumor in the prostatectomy specimen after neoadjuvant therapy.

SECONDARY OUTCOMES:
Residual cellularity rate | 3 months
  To compare the rate of residual cellularity ≤ 30% in the prostatectomy specimen after neoadjuvant therapy.
Pathologic downgrading | 3 months
  To compare the rate of pathologic downgrading to ≤ ypT2N0 in the prostatectomy specimen after neoadjuvant therapy.
PSA decline rate | 3 months
  To compare the rate of PSA decline ≥ 50% and 90% after 3 months of neoadjuvant therapy.
Rate of positive surgical margins | 3 months
  To compare the rate of positive surgical margins in the prostatectomy specimen after neoadjuvant therapy.
Rate of undetectable PSA | 12 months
  To compare the rate of patients with undetectable PSA 12 months after radical prostatectomy.
Rate of Grade ≥ 3 CTCAE adverse events | 3 months
  To compare the rate of CTCAE grade 3 or higher adverse events of the neoadjuvant therapy arms

OTHER OUTCOMES:
Rate of Magnetic Resonance Image Downstaging after Neoadjuvant Therapy | 3 months
  To compare the MR image downstaging after neoadjuvant therapy with pathologic analysis of the prostatectomy specimen
Exploratory analysis to correlate tissue expression of PSA, CYP17, Ki67, and AR with pathologic response. | 3 months
  To correlate the expression of PSA, CYP17, Ki67, and AR by immunohistochemistry with pCR/npCR in the prostatectomy specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Diogo A Bastos, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No